CLINICAL TRIAL: NCT06362135
Title: The Evaluation of the Effectiveness of Virtual Home Visits for Stroke Patients and Their Caregivers as Part of Home Health Services.
Brief Title: Virtual Home Visits for Stroke Patients and Their Caregivers
Acronym: INHABASAEV
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The Scientific and Technological Research Council of Turkey (Other)
Responsible Party: Principal Investigator, Yasemin Demir, Dr. (Assistant professor), Akdeniz University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 0733
Record Dates: First submitted 2024-04-08; First posted 2024-04-12 (Actual); Last update posted 2024-04-15 (Actual); Status verified 2024-04

CONDITIONS: Stroke; Caregiver; Virtual; Home Visit
MeSH Terms: conditions — Stroke | interventions — Control Groups

STUDY DESIGN:
Intervention Model Description: Parallel Assignment Virtual visit with stroke patient and their caregiver
Who Masked: Outcomes Assessor
Masking Description: Telephone support or virtual meeting during the research process will be provided by an independent interviewer.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Virtual home visit (Experimental): to evaluate the effectiveness of virtual home visits in terms of time, cost and caregiver competence
  Interventions: Device: Virtual Home Visit
- Home visit (Active Comparator): to evaluate the effectiveness of home visits in terms of time, cost and caregiver competence
  Interventions: Device: Control Group

INTERVENTIONS:
Device: Virtual Home Visit — The virtual home visit will be made through the mobile application developed by the researchers. First, the patients who meet the sampling criteria will be included in the study after the caregivers of the patients apply to the Antalya Health Directorate Antalya Training and Research Hospital Home Health Unit. The virtual home visit is scheduled twice
  Arms: Virtual home visit
Device: Control Group — "Face-to-face home visits will be carried out by the Antalya Education and Research Hospital home health team, as planned.
  Other Names: Home visit
  Arms: Home visit

SUMMARY:
The primary aim of this study is to evaluate the effectiveness of virtual home care for stroke patients and their caregivers. The secondary purpose is to evaluate the usability of the application by developing a mobile application for use in virtual home visits.

The study will be carried out using the mixed research model, in which quantitative and qualitative methods are used together. The population of the research will consist of patients and caregivers with the diagnosis of hemorrhage, infarction, cerebrovascular accident and cerebral infarction, who applied to the Antalya Provincial Health Directorate Antalya Training and Research Hospital Home Health Unit, where the study is planned to be conducted. The sample of the study will consist of stroke patients and caregivers who meet the criteria for inclusion in the study. The first phase of the study was designed as a parallel group, single center and single blind randomized controlled trial to evaluate the effectiveness of virtual home visits in terms of time, cost and caregiver competence. The experimental group was the patient/patient relative group who made a virtual home visit, the control group will consist of 48 patients/patient relatives who have been visited face-to-face. In the second phase of the study, semi-structured interview method will be used to determine the views of patients/patient relatives about virtual home visits. In order to evaluate the usability of the developed application, a usability survey will be applied to the group that has visited the virtual home.

With the results of this study, telemedicine applications in home care services will help to increase accessibility to home care services and reduce health care costs.considered to contribute. At the same time, it is expected that the results of the study will contribute to the scientific literature in the field of design and application of telemedicine services, which are developing and spreading

DETAILED DESCRIPTION:
Stroke is one of the leading causes of death in our country, with 22.2%. In addition, stroke, the most common disease diagnosis, has a prevalence of 35%. Treatment of this disease begins in the hospital and continues at home. Treatment and spread over many years. There are barriers due to reasons such as the inability of stroke patients to come to the outpatient clinic, bed dependency, old age, and living outside the central district due to the lack of advanced specialist areas related to stroke in the center and big cities. In addition, the Covid-19 pandemic has made it difficult for the stroke patient to benefit from home health care. In our country, home care services are generally for conical diseases. One of the chronic diseases in the first three of these is stroke patients, whose medical diagnosis is called cerebrovascular disease. Stroke patients constitute an important part of home care services.

Remote healthcare provides many advantages to healthcare professionals and patients with chronic disease diagnosis. Some of these advantages are; TÜSEB Home Health Services Report (2021) states that virtual home visits are used to reduce the risk of transmission of Covid-19 disease during the pandemic. In addition to the many advantages of remote health services, problems such as users' readiness, usability, technology literacy, attitudes, internet access while using remote health services still continue today.

ELIGIBILITY:
Inclusion Criteria:

* Being willing to participate in the study,
* Hospitalization with the diagnosis of (stroke, hemorrhage, infarction, cerebrovascular accident and cerebral infarction),
* Districts of Antalya Training and Research Hospital
* The patient's * Barthel Activities of Daily Living Index dependency level is complete, severe, moderate, and mildly dependent.
* For pressure ulcer risk **Braden Risk Assessment Tool
* For caregivers;
* Having internet access Being primarily responsible for the care of the patient (who performs the daily activities of the patient during the intervention),
* The caregiver has internet access,
* At least one person in the house where the patient lives is using the internet,
* In the case of more than one caregiver, the most willing caregiver,

Exclusion Criteria:

* The lack of volunteerism of the stroke patient and family
* The patient has a history of addiction other than stroke,
* Caregiver not having internet access
* Caring for a fee,

Unfollowing Criteria

* Patient's death
* Patient and caregiver wanting to quit the study

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Estimated)
Dates: Start 2023-08-01 (Actual); Primary Completion 2024-12-01 (Estimated); Study Completion 2025-03-01 (Estimated)

PRIMARY OUTCOMES:
Effect of Virtual and Face to face to home visit | Change from baseline effect of visit at 0,3 month
  For virtual and face-to-face visits, it includes the type of visit, the health personnel who made the visit, the number of visits, the average visit time (minutes), the duration of the home visit (in terms of time and distance), the materials used in the home visit. It will also be created to calculate the cost effective.
Level of competence of stroke caregiver | Change from baseline effect of virtual visit at 0, 3 month (minimum 4 points, maximum 16 points)
  Caregiver Competence Scale Caregiver Competence Scale
Frequency of unplanned hospital readmission | Change from baseline effect of virtual visit at 3 month
  Unplanned admission to hospital after discharge: The content of the form includes questions about hospital applications after discharge and the reasons for application.

SECONDARY OUTCOMES:
Effect of the virtual home visit | Change from baseline effect of virtual visit at 3 month (A score ranging from 0-100 is obtained from the scale. A higher score indicates an increased level of usability).
  System Usability Scale

CONTACTS AND LOCATIONS:
Locations (1):
- Yasemin Demi̇r Avci̇, Antalya, Turkey (Türkiye)